CLINICAL TRIAL: NCT05553795
Title: Drainless Robot-assisted Minimally Invasive Esophagectomy
Acronym: RESPECT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Following a safety analysis and assessment of the complications encountered by external experts, it was decided to terminate recruitment prematurely
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VTG-11
Record Dates: First submitted 2022-08-19; First posted 2022-09-23 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
Keywords: Esophagectomy; Enhanced Recovery after Surgery (ERAS); Robot-assisted minimally invasive esophagectomy (RAMIE)
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chest Tubes

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicentric trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A - Early removal of chest drain (Experimental)
  Interventions: Procedure: Early removal of chest drain
- B - Control (Other)
  Interventions: Procedure: Chest drain

INTERVENTIONS:
Procedure: Early removal of chest drain — Chest drains are removed 3 hours after the end of surgery in absence of contraindications in arm A.
  Arms: A - Early removal of chest drain
Procedure: Chest drain — The chest drains in arm B are removed during the further postoperative course according to standard algorithm.
  Arms: B - Control

SUMMARY:
The aim of this study is the evaluation of two different chest drain management strategies in patients undergoing robot-assisted minimally invasive esophagectomy (RAMIE) for esophageal cancer with regard to perioperative complications until discharge.The primary objective of the study is to investigate whether the intensity of postoperative pain can be significantly reduced by avoiding thoracic drains after RAMIE. We assume that this will influence secondary endpoints such as early recovery and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective RAMIE for esophageal cancer with intrathoracic esophagogastrostomy (Ivor-Lewis)
* American Society of Anesthesiologists (ASA) score ≤ III
* Eastern Cooperative of Oncology Group (ECOG) status ≤ II
* Patient suitable for both surgical techniques
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent

Exclusion Criteria:

* Open esophagectomy (either abdominal or during the thoracic part)
* Emergency operations
* ASA IV
* ECOG > II
* Chronic pain syndromes requiring routine analgesics
* Simultaneous lung resection
* Presence of contraindications to the use of epidural anesthesia (e.g. coagulopathies, anticoagulation or allergies)
* Participation in an interventional trial, which interferes with the outcome
* Impaired mental state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Day 2 after surgery
  Postoperative pain according to a numeric rating scale

SECONDARY OUTCOMES:
Mean postoperative pain | Day 4 after surgery
  Postoperative pain according to a numeric rating scale
Additional analgesic drug use | Day 4 after surgery
  opioids [mg], non-opioids [mg]
Postoperative mobilization | Day 7 after surgery
  steps per day as measured with an activity tracker
Postoperative morbidity | Through hospital stay, an average of 14 days
  The postoperative morbidity of all patients is assessed with the comprehensive complication index based on Clavien Dindo classification from postoperative day 1 until day of discharge
Postoperative mortality | Through hospital stay, an average of 14 days
  The postoperative mortality of all patients is assessed between operation date and date of death of any cause during hospital stay
Daily postoperative pain | Day 7 after surgery
  Postoperative pain according to a numeric rating scale measured daily from postoperative day 1-7

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Kirchberg, Dr. med., Principal Investigator — Department of Gastrointestinal-, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus
Locations (1):
- Department of Gastrointestinal-, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mussle B, Kirchberg J, Buck N, Radulova-Mauersberger O, Stange D, Richter T, Muller-Stich B, Klotz R, Larmann J, Korn S, Klimova A, Grahlert X, Trips E, Weitz J, Welsch T. Drainless robot-assisted minimally invasive oesophagectomy-randomized controlled trial (RESPECT). Trials. 2023 May 2;24(1):303. doi: 10.1186/s13063-023-07233-z. PMID 37127683